CLINICAL TRIAL: NCT03355924
Title: DMEK And Cataract Surgery: Comparison Of Sequential Versus Combined Procedure
Acronym: CISIPHE
Status: Completed | Type: Observational
Sponsor: Centre Hospitalier Régional Metz-Thionville (Other)
Responsible Party: Sponsor
Other Study IDs: 2016-08Obs-CHRMT
Record Dates: First submitted 2017-11-23; First posted 2017-11-28 (Actual); Last update posted 2023-08-24 (Actual); Status verified 2017-11

CONDITIONS: Cataract; Corneal Graft
MeSH Terms: conditions — Cataract

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The aim of this study is to describe the outcomes of phaco-DMEK (Descemet Membrane Endothelial Keratoplasty ) according to a sequential versus a combined procedure

DETAILED DESCRIPTION:
The study included patients who underwent DMEK combined or not with cataract surgery between January 2014 and march 2016. Were excluded patients with other ocular comorbidity, and those who had graft after a first graft failure. The main outcome was BVCA measured at one year. The post-operative follow up was down at D7, M1, M3, M6, and M12. Secondary outcomes were; the mean time to visual recovery and influence of the delay between cataract removal and DMEK.

ELIGIBILITY:
Inclusion Criteria:

* patients who underwent DMEK combined or not with cataract surgery

Exclusion Criteria:

* patients with other ocular comorbidity, and those who had graft after a first graft failure

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: patients who underwent DMEK combined or not with cataract surgery
Sampling Method: Non-Probability Sample
Enrollment: 31 (Actual)
Dates: Start 2016-11-01 (Actual); Primary Completion 2017-05-30 (Actual); Study Completion 2017-05-30 (Actual)

PRIMARY OUTCOMES:
Best visual acuity | Month 12
  logMar